CLINICAL TRIAL: NCT06339983
Title: Comparative Effects of Manual Scar Mobilization Versus Myofascial Cupping Technique on Pain, Physical Characteristics, and Appearance of the Cesarean Scar
Brief Title: Effects of Scar Mobilization Versus Myofascial Cupping Technique on Cesarean Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0566
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Section; Complications, Wound, Hematoma
Keywords: Cesarean Scar; Mobilization; Manual therapy
MeSH Terms: conditions — Wounds and Injuries; Hematoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Scar Mobilization: (Experimental): Group will undergo manual scar mobilization therapy. In this therapy, deep pressure on some point of the area of the scar will be given which will be perpendicular to the skin which will be followed by skin rolling. The manual therapy will include different techniques such as rolling, stroking, superficial rubbing, deep rubbing, breaking up, and pinching. The therapy will continue for 15 minutes.
  Interventions: Other: Manual Scar Mobilization Therapy:
- Myofascial Cupping Therapy (Active Comparator): Group will receive myofascial cupping therapy. In this method, the patient will lie down on the bed with an exposed scar area. Application areas will be cleaned and herbal oil or cream will be applied. A disposable plastic cup (5cm) will be positioned at THE selected area of the cesarean scar. Then, negative pressure will be applied using a mechanical vacuum pump, the cup will be gently slid around the selected area rhythmically to get a massage-like effect for approximately 5-15 minutes. Then the cup will be removed gently. After this, the application areas will be cleaned.
  Interventions: Other: Myofascial Cupping Therapy:

INTERVENTIONS:
Other: Manual Scar Mobilization Therapy: — In this therapy, deep pressure on some point of the area of the scar will be given which will be perpendicular to the skin and will be followed by skin rolling
  Arms: Manual Scar Mobilization:
Other: Myofascial Cupping Therapy: — A disposable plastic cup (5cm) will be positioned at THE selected area of the cesarean scar. Then, negative pressure will be applied using a mechanical vacuum pump, the cup will be gently slid around the selected area rhythmically to get a massage-like effect
  Arms: Myofascial Cupping Therapy

SUMMARY:
Study focuses on comparing the effects of manual scar mobilization and myofascial cupping techniques on the outcomes of pain, physical characteristics, and appearance of cesarean scars. The study aims to contribute valuable insights into tailored interventions for improving cesarean scars. The randomized clinical trial will involve 52 participants, primigravida women aged 20 to 40 with completely healed but painful cesarean scars. Excluding those with previous scar therapy or infectious scars, the participants will be divided into two groups, with Group A receiving manual scar mobilization therapy and Group B receiving myofascial cupping therapy, both administered twice a week for four weeks. Pain assessment will be conducted using a numeric pain rating scale (NPRS), while physical characteristics and appearance will be evaluated using the Manchester Scar Scale for cesarean scars (MSS). The data collected will be analyzed using SPSS version 29.

DETAILED DESCRIPTION:
A cesarean is a surgical procedure used to deliver a baby through an incision in the mother's abdomen and uterus. Manual scar mobilization and myofascial cupping techniques are some of the beneficial techniques to treat the scar. The research aims to understand the comparative effects of both techniques to know the potential benefits of these techniques on the outcome of pain, physical characteristics, and appearance of the cesarean scar. This study contributes valuable insights into comparing tailored interventions for improving the cesarean scar. This will be a randomized clinical trial conducted on 52 participants. Data will be collected from KulsoomShoukat Medical Complex, Faisalabad by using a non-probability convenience sampling technique. Primigravida women aged from 20 to 40 who have 6 months post cesarean completely healed but painful scars and who haven't undergone any scar therapy before will be included in the study. On the contrary, participants with any previous scar therapy or having infectious scars will be excluded from the study. A sample of 48 will be divided into 2 groups through random allocation. Group A will undergo manual scar mobilization therapy for 15 minutes on a cesarean scar twice a week. Group B will receive myofascial cupping therapy for 15 minutes twice a week. Treatment in both groups will be given for 4 weeks and pain will be assessed before 4 weeks and then after 4 weeks by a numeric pain rating scale (NPRS). Physical characteristics and appearance will be assessed by the Manchester Scar Scale for cesarean scar (MSS) in both groups pre and post-intervention. Data will be analyzed using SPSS version 29.

ELIGIBILITY:
Inclusion Criteria:

* Women with Pfannenstiel Cesarean section scar
* Primigravida
* Women who didn't undergo any scar therapy
* The age of the scar should be under 6 months
* Women with a completely healed scar
* Women with painful scar

Exclusion Criteria:

* Diabetic women
* Skin irritation or infection at the scar site
* Women with Diastasis Recti Abdominis
* Obese women (BMI<35%)
* Women with Hysterectomy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 4 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes.
Manchester Scar Scale (MSS) | up to 4 weeks
  In 1998 Beausang et al proposed a scale to assess scars which is the Manchester Scar Scale (MSS). It rates the different physical characteristics of scar which are contour to surrounding skin (range from flush to keloid) and texture (range normal to hard). Scores from the parameters are then all together to get the total score, with higher scores representing clinically worse scars. Manchester scar scale also gives the appearance of the scar that is color (from perfect to mismatched), relationship with the surrounding skin (shiny or mate), and distortion (none to severe). Then the score is added to get the overall opinion about the scar.

CONTACTS AND LOCATIONS:
Overall Officials: Kainat Ashfaq, MS*, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Kulsoom Shoukat Medical Complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbas F, Ud Din RA, Sadiq M. Prevalence and determinants of Caesarean delivery in Punjab, Pakistan. East Mediterr Health J. 2019 Jan 23;24(11):1058-1065. doi: 10.26719/2018.24.11.1058. PMID 30701520
- [Background] Singh N, Pradeep Y, Jauhari S. Indications and Determinants of Cesarean Section: A Cross-Sectional Study. Int J Appl Basic Med Res. 2020 Oct-Dec;10(4):280-285. doi: 10.4103/ijabmr.IJABMR_3_20. Epub 2020 Oct 7. PMID 33376704
- [Background] Vejnovic TR. [Cesarean delivery--Vejnovic modification]. Srp Arh Celok Lek. 2008 May;136 Suppl 2:109-15. doi: 10.2298/sarh08s2109v. Serbian. PMID 18924480
- [Background] Olszewska K, Ptak A, Rusak A, Debiec-Bak A, Stefanska M. Changes in the scar tissue structure after cesarean section as a result of manual therapy. Adv Clin Exp Med. 2024 Apr;33(4):387-395. doi: 10.17219/acem/169236. PMID 37665082
- [Background] Gilbert I, Gaudreault N, Gaboury I. Exploring the Effects of Standardized Soft Tissue Mobilization on the Viscoelastic Properties, Pressure Pain Thresholds, and Tactile Pressure Thresholds of the Cesarean Section Scar. J Integr Complement Med. 2022 Apr;28(4):355-362. doi: 10.1089/jicm.2021.0178. Epub 2022 Jan 13. PMID 35426735
- [Background] Lubczynska A, Garncarczyk A, Wcislo-Dziadecka D. Effectiveness of various methods of manual scar therapy. Skin Res Technol. 2023 Mar;29(3):e13272. doi: 10.1111/srt.13272. PMID 36973982
- [Background] Pianese L, Bordoni B. The Use of Instrument-Assisted Soft-Tissue Mobilization for Manual Medicine: Aiding Hand Health in Clinical Practice. Cureus. 2022 Aug 31;14(8):e28623. doi: 10.7759/cureus.28623. eCollection 2022 Aug. PMID 36059328